CLINICAL TRIAL: NCT05581329
Title: Change in Skin Surface Temperature at the Neck When Using Acupuncture at Houxi Point in Healthy Volunteers: a Randomized Controlled Trial
Brief Title: Change in Skin Surface Temperature at the Neck When Using Acupuncture at Houxi Point in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bui Pham Minh Man (Other)
Responsible Party: Sponsor-Investigator, Bui Pham Minh Man, Medical Doctor, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 679/HDDD-DHYD
Record Dates: First submitted 2022-10-10; First posted 2022-10-14 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
Keywords: Acupuncture; Skin surface temperature
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: 2-arm parallel design, randomized, controlled and single blinded trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: acupoints on the left hand (Experimental): Participants will be received acupuncture at the control acupoint (Yuji - LU10) in the first trial phase, and the second trial phase will be conducted after 07 days at the research acupoint (Houxi - SI3). In each time, skin surface temperature at the neck area will be recorded.
  Interventions: Procedure: Acupuncture
- Group B: acupoints on the right hand (Experimental): Participants will be received acupuncture at the control acupoint (Yuji - LU10) in the first trial phase, and the second trial phase will be conducted after 07 days at the research acupoint (Houxi - SI3). In each time, skin surface temperature at the neck area will be recorded.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture is a method of inserting very thin needles into special points on the body which are called acupoints. To conduct this intervention, we will use disposable acupuncture needles the size of 0.30 x 13 mm to acupuncture the control acupoint (Yuji - LU10) in the first session and the research acupoint (Houxi - SI3) in the second session.

SUMMARY:
Acupuncture is a method of inserting very thin needles into special points on the body which are called acupoints, to treat diseases. This treatment has been widely applied in health care for over 2500 years. Currently, by synthesizing the results of many clinical studies, the World Health Organization (WHO) has recognized the importance of acupuncture as an effective treatment for various diseases. However, the specific effect of acupoints is still controversial. Until now, several studies have shown that acupoints are associated with certain areas of the human body that are far from the acupoints and can alter the temperature of those area. In our study, we will survey on the change in skin surface temperature at the neck when using acupuncture at Houxi point in healthy volunteers.

DETAILED DESCRIPTION:
Participants and Methods: A randomize controlled trial will be conducted by comparing the change in the skin surface temperature before and after using acupunture at the control acupoint (Yuji - LU10) and the research acupoint (Houxi - SI3) on either the left or right hand in healthy volunteers. A total of 60 participants will be randomly assigned to 2 group (A and B) and the allocation was 1:1. Both groups will undergo two trial phases 07 days apart, corresponding to one acupoint on the same hand in each step. Group A (acupoints on the left hand): participants will be received acupuncture at the control acupoint (Yuji - LU10) in the first trial phase, and the second phase will be conducted after 07 days at the research acupoint (Houxi - SI3). Group B: proceeding similarly to group A, but the points are on the right hand. The primary outcome will be the change in skin surface temperature at the neck when using acupuncture at Houxi point on each hand. This trial will be performed as a 2-arm parallel design, randomize, controlled and single blinded.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females were individual age between enough 18 and 30 years old.
* BMI: 18.5 - 23 kg/m2
* Mental alertness, good contact, cooperation with researchers.
* Having no psychiatric stress problem during acupuncture day (confirmed by answering the DASS21 questionnaire with stress point less than 15 points).
* Vital sign within normal limits:

  * Heart rates from from 60 to 99 beats/minute.
  * Systolic blood pressure between 90 and 139 mmHg.
  * Diastolic blood pressure between 60 and 89 mmHg.
  * Body temperature: 36.59 ± 0.43 0C.
  * Breathing rate: 16 ± 3 respirations/minute .
* Having no disease or using drugs that change the body temperature.
* Not currently participating in other intervention studies.
* Volunteers who agree to participate and sign the Informed Consent Form, following a detailed explanation of clinical trials.
* Having no acupuncture knowledge and experience yet.

Exclusion Criteria:

* Playing sport 2 hours before the study.
* Taking stimulant (alcohol, beer, coffee and tobacco) within 24 hours before conducting the study.
* Staying up late at night or having insomnia before the day of the study.
* Women who were in menstruation period, pregnancy, or breastfeeding.
* Having skin injuries, dermatitis-skin infections or wounds in the area to be investigated.
* Curently having neck-pain or other diseases that could affect or interfere with outcomes, including common cold.
* Currently taking sedatives or drugs that cause vasodilation, affect blood pressure and heart rate.
* Applying chemical or pharmaceutical products to the site of the skin to be investigated before conducting the study.
* Using physical therapy, heat therapy, cupping therapy, massage, acupuncture in the site of the skin to be investigated within 24 hours.
* Anxiety, depression, stress before conducting the study with DASS 21 score < 15.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The change in skin surface temperature at the neck when using acupuncture at Houxi point on each hand. | During procedure
Survey the change in temperature at the neck area respectively when using acupuncture at the left and right research acupoints (Houxi - SI3) compared with the control acupoints group (Yuji - LU10). | During procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Traditional medicine - University of Medicine and Pharmacy of Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Demographic characteristic and outcome data will be shared
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- See also: Mo MJ, Hwang DR, Lee JH, et al. Analysis on the Acupuncture Contents of the Domestic Neck Pain and HIVD-Cervical Spine Clinical Studies: a literature review. 2017;34(2):113-125. — https://www.semanticscholar.org/paper/Analysis-on-the-Acupuncture-Contents-of-the-Neck-a-Mo-Hwang/1da4e93815c93ce47e946b21a3d4b9d566105252
- See also: Guan L, Li G, Yang Y, Deng X, Cai PJNRR. Infrared thermography and meridian-effect evidence and explanation in Bell's palsy patients treated by moxibustion at the Hegu (LI4) acupoint: Overall regulation or a specific target?. 2012;7(9):680. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4347008/
- See also: Ots T, Kandirian A, Szilagyi I, DiGiacomo SM. The selection of dermatomes for sham (placebo) acupuncture points is relevant for the outcome of acupuncture studies: a systematic review of sham (placebo)-controlled randomized acupunc — https://pubmed.ncbi.nlm.nih.gov/32026725/
- See also: Molsberger A, Manickavasagan J, Abholz H, Maixner W, Endres HJEJoP. Acupuncture points are large fields: the fuzziness of acupuncture point localization by doctors in practice. 2012;16(9):1264-1270. — https://pubmed.ncbi.nlm.nih.gov/22492604/